CLINICAL TRIAL: NCT05430100
Title: The Effect of usıng Breast mılk pacıfıer, Sucrose pacıfıer and pacıfıer ın reducıng the paın That Occurs durıng orogastrıc Tube ınsertıon ın Preterm Newborns
Brief Title: Reducing Pain During Orogastric Tube Placement in Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Dilek Konukbay, Assistant professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBU-KONUKBAY-002
Record Dates: First submitted 2022-05-31; First posted 2022-06-24 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Preterm; Pain; Nursing Caries
Keywords: Pain; preterm; orogastric tube; Neonatal Intensive Care Unit
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Intervention Model Description: A total of 4 groups will be involved in our research. These are; - Breast milk pacifiers group, - Sucrose pacifiers group, - Pacifiers group, - Control group. The numbers to be given to the groups will be determined by lot method. In the research, the assignment of the participants to the groups will be made using the "block randomization method". Randomization will be provided by the researcher using microsoft excel. By typing the numbers from 1 to 100 in cell A, adding the RAND() operation to cell B, the number will be generated in all rows from 1 to 100. Then, the sorting process will be performed on the numbers in cell B and a random list will be created in column A. After evaluating the inclusion criteria and obtaining consent from the participants, it will be determined which group the preterm newborn will be in.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breast Milk Pacifiers Group (Experimental): To determine the effectiveness of breast milk pacifier in reducing pain caused by Orogastric Tube (OGT) insertion in preterm newborns by monitoring behavioral and physiological changes in infants.
  Interventions: Other: The effect of usıng breast mılk pacıfıer ın reducıng the paın that occurs durıng orogastrıc tube ınsertıon ın preterm newborns
- Sucrose Pacifiers Group (Experimental): To determine the effectiveness of sucrose pacifier in reducing pain caused by Orogastric Tube (OGT) insertion in preterm newborns by monitoring behavioral and physiological changes in infants.
  Interventions: Other: The effect of usıng sucrose pacıfıer ın reducıng the paın that occurs durıng orogastrıc tube ınsertıon ın preterm newborns
- Pacifiers Group (Experimental): To determine the effectiveness of pacifier in reducing pain caused by Orogastric Tube (OGT) insertion in preterm newborns by monitoring behavioral and physiological changes in infants.
  Interventions: Other: The effect of usıng pacıfıer ın reducıng the paın that occurs durıng orogastrıc tube ınsertıon ın preterm newborns
- Control Group (No Intervention): The camera recording will be started 5 minutes before the OGT insertion procedure and the routine OGT placement process will be performed. No pain-related procedures are performed during routine OGT in the NICU.

INTERVENTIONS:
Other: The effect of usıng breast mılk pacıfıer ın reducıng the paın that occurs durıng orogastrıc tube ınsertıon ın preterm newborns — 5 Minutes before the OGT insertion, the camera recording will be started and the preterm newborn will be given a breast milk pacifier. After the breast milk pacifier in the OGT intervention group is placed in the mouth as a leak from the edge of the given baby's mouth, the baby's esophagus will be placed by advancing from there to the stomach with the swallowing reflex. It will be checked whether the OGT is in the right place. Registration will be stopped after the evaluation period is completed and the baby is provided with comfort. But the recording will continue so that there are no time restrictions for tracking the crying time of the baby who continues to cry during placement. In terms of the reliability of the research results, nothing should be given orally to a preterm newborn at least 30 minutes before the procedure.
  Other Names: Sucrose Pacifiers Group; Pacifiers Group
  Arms: Breast Milk Pacifiers Group
Other: The effect of usıng sucrose pacıfıer ın reducıng the paın that occurs durıng orogastrıc tube ınsertıon ın preterm newborns — The camera recording will be started 5 minutes before the OGT insertion procedure and the newborn will be given a sucrose-sweetened pacifier. After the sucrose-sweetened pacifier in the OGT intervention group is placed in the mouth as a leak from the edge of the given baby's mouth, the baby's esophagus will be placed by advancing from there to the stomach with a swallowing reflex. It will be checked whether the OGT is in the right place. Registration will be stopped after the evaluation period is completed and the baby is provided with comfort. But the recording will be continued so that there are no time restrictions for tracking the crying time of the baby who continues to cry during placement. In terms of the reliability of the research results, nothing should be given orally to a preterm newborn at least 30 minutes before the procedure.
  Other Names: Breast Milk Pacifiers Group; Pacifiers Group
  Arms: Sucrose Pacifiers Group
Other: The effect of usıng pacıfıer ın reducıng the paın that occurs durıng orogastrıc tube ınsertıon ın preterm newborns — The camera recording will be started 5 minutes before the OGT insertion procedure and the newborn will be given a pacifier. After the pacifier in the OGT intervention group is placed in the mouth as a leak from the edge of the given baby's mouth, the baby's swallowing reflex will be placed by moving the esophagus from there to the stomach. It will be checked whether the OGT is in the right place. Registration will be stopped after the evaluation period is completed and the baby is provided with comfort. But the recording will be continued so that there are no time restrictions for tracking the crying time of the baby who continues to cry during placement.
  Other Names: Breast Milk Pacifiers Group; Sucrose Pacifiers Group
  Arms: Pacifiers Group

SUMMARY:
The aim of this study is to determine the effectiveness of 3 different methods (breast milk pacifier, sucrose pacifier and pacifier) in reducing pain caused by Orogastric Tube (OGT) insertion in preterm newborns by monitoring behavioral and physiological changes in infants. The study was planned as a randomized controlled experimental study.

DETAILED DESCRIPTION:
Babies born before the 37th week of pregnancy are defined as preterm. Preterm newborns need Neonatal Intensive Care Unit (NICU) due to their immature characteristics. NICU includes many diagnostic and therapeutic procedures associated with pain. Babies are exposed to many painful procedures during their stay in the NICU. The International Association for the Study of Pain (IASP) defines pain as "an uncomfortable sensory and emotional experience that develops as a result of existing or potential tissue damage or is described by this damage".

It is known that pain begins to be felt by the fetus from the intrauterine second trimester. Especially, preterm newborns are more vulnerable to the effects of pain exposure due to their developing central and peripheral nervous systems and are more sensitive to pain due to low pain thresholds. Therefore, developing appropriate pain control strategies, especially for preterm newborns, is both a medical and ethical responsibility. In their study, Zhao et al. defined pain as a complex and multidimensional phenomenon experienced in the NICU for preterm newborns. In a study by Mooney-Leber et al. with 430 newborns, it was stated that approximately 80 painful procedures were performed without specific analgesia. Reducing the pain of term and preterm newborns experiencing pain with effective and safe methods is a fundamental right of all newborns.

The sucking reflex in preterm newborns is 28th in intrauterine life. it begins to develop after 32-34 weeks of gestation. during the gestational week, sucking and swallowing reflexes develop. Preterm newborns admitted to NICU are fed through the orogastric tube (OGT) until they can coordinate their sucking, swallowing, and breathing. A probe inserted through the mouth into the esophagus (esophagus) and from there into the stomach is called an orogastric tube. Measurement of OGT placement in preterm newborns; it is made in such a way that it comes from the baby's earlobe to the middle line of the mouth, and from there to the middle line between the Deciphoid protrusion and the umbilical cord. Taking the black markers on the probe as reference points, the length of the probe is adjusted accordingly, the tip should not be touched so that the tip of the probe is not contaminated. The process is stopped when the OGT reaches the point measured before the operation. The stomach contents are checked. OGT is detected at the edge of the mouth when it is sure of its location.

The placement and use of OGT is one of the most common nursing practices applied as a therapeutic and diagnostic method in NICU . It is used for enteral nutrition, drug administration, drainage of the contents of the stomach/small intestine or for decompression and gastric analysis in hospitalized infants. However, OGT placement is a painful, stressful and troublesome procedure for preterm newborns. In preterm newborns, OGT placement is performed frequently until the development of the sucking and swallowing reflex is completed. The fact that the pain is felt intensely, the application is frequent, causes more pain in preterm newborns. It has been stated that recurrent pain leads to decreased brain oxygenation, causing excitotoxic damage to the developing neurons of newborn babies, increasing anxiety, changing sensitivity to pain, stress-related diseases, hyperactivity, attention deficit and may have negative effects on the development of social abilities.

Atraumatic care, which is included in nursing approaches, is defined as therapeutic care or interventions that eliminate or minimize physical stress factors. In line with atraumatic nursing care, pain management is considered as a basic element of care. Newborn nurses closely testify to pain and stress. For the prevention of pain, it is important to provide individual and holistic nursing care. Accordingly, the knowledge of pharmacological and non-pharmacological methods in the management of pain by the nurse has a positive effect on the evaluation of pain in infants and pain management. The use of non-pharmacological methods that are easy to apply and low in cost by neonatal nurses is important for effective pain management. Non-pharmacological methods; sucking, sucrose or dextrose, breastfeeding (breast milk), kangaroo care (skin-to-skin contact), wrapping, massage, touching the face, positioning (fetal position), acupuncture and music therapy can be listed as non-nutritious or nutritious. When the literature is examined, it is stated that it is more effective to use more than one non-pharmacological method together in the use of non-pharmacological methods instead of their use alone . Given the frequency of OGT administration and the sensitivity of preterm infants, ensuring the management of pain during the OGT process will positively affect the development of the preterm baby. There are studies in the literature that different non-pharmacological methods used in OGT placement are effective in reducing pain in preterm newborns. In this study, a study planned in which the methods of using breast milk pacifiers, sucrose pacifiers, and pacifiers were compared together to reduce the pain caused by orogastric tube insertion in preterm newborns was not found in the literature.

The use of a pacifier (non-nutritious suction), one of the non-pharmacological methods included in the scope of the study, is used in routine practice to improve the ability to suck in preterm newborns. To stimulate sucking in non-nutritious sucking, a warning is given by touching the cheek, lips, tongue, gums, jaw and palate. The purpose of this method is to strengthen sucking by stimulating the oral motor functions of the preterm baby. In this way, coordination between sucking, swallowing and during respiration is supported. It is stated that sucrose, which will be used as another method, is effective in reducing pain in some studies, but there may be problems in terms of cost and access in routine applications. Breast milk is a miraculous food that meets all the needs of the newborn in terms of the components it contains, and it has the property of preventing the transmission of pain sensation by stimulating opioids with the nutrients it contains and blocking the pain fibers. It is evaluated that determining the effects on pain management by comparing the pacifier, breast milk pacifier and sucrose pacifier methods in reducing the pain that will occur during the OGT insertion procedure in preterm newborns, the outcomes will contribute to the literature by guiding the effective pain management during the OGT procedure in preterm newborns hospitalized in the NICU.

Hypotheses Of The Study:

In reducing the pain caused by OGT insertion in preterm infants, Hypothesis 0 (H0): There is no difference between breast mılk pacıfıers, sucrose pacıfıers and pacıfıers methods.

Hypothesis 1.1 (H1.1): The breast mılk pacıfıers method is more effective than the control group.

Hypothesis 1.2 (H1.2): The sucrose pacıfıers method is more effective than the control group.

Hypothesis 1.3 (h.1.3): The pacifier method is more effective than the control group.

Hypothesis 1.4 (H1.4): The breast milk pacifier method is more effective than the sucrose pacifier group.

Hypothesis 1.5 (H1.5): The breast milk pacifier method is more effective than the pacifier group.

Hypothesis 1.6 (H1.6): The sucrose pacıfıers method is more effective than breast milk pacifier group.

Hypothesis 1.7 (H1.7): The sucrose pacıfıers method is more effective than pacifier group.

Hypothesis 1.8 (H1.8): The pacifier method is more effective than the breast milk pacifier group.

Hypothesis 1.9 (H1.9): The pacifier method is more effective than the sucrose pacifier group.

Place And Tıme Of The Study:

The study was planned to be carried out after the necessary ethics committee permissions were obtained from the Human Research Ethics Committee of Ankara University Faculty of Medicine. July 2022- july 2023 will be conducted at Ankara University Neonatal Intensive Care Unit. There are 30 nurses in the Neonatal Intensive Care Unit and 4. It serves up to the step.

Unıverse And Sample Of The Study:

In the analysis of the research hypotheses, it is planned to perform analyzes of two and more than two group comparisons and the highest sample size calculated according to the statistical method to be performed is taken as the basis. In this study, "G. Using the "Power-3.1.9.2" program, the sample size was calculated to compare multiple 3 or more groups at a 95% confidence level. As a result of the analysis, α=0.05, the standardized effect size was taken as 0.460461 (high grade) using a similar study conducted in this field earlier, and the minimum sample volume was calculated as 56 with a theoretical strength of 0.80.

ELIGIBILITY:
Inclusion Criteria:

* A gestational age of 30-34 weeks ,
* Having his mother's milk
* Stable state of health
* The fact that the preterm baby has not previously had an orogastic tube inserted
* Having spontaneous breathing
* Being fed through the orogastric tube
* Not taking opioids or non-opioid analgesics
* He did not receive a painful stimulus until 30 minutes before the intervention,
* Volunteer consent of the parents of the preterm neonate to participate in the study

Exclusion Criteria:

* Have any congenital abnormalities on the face or oral cavity,
* The need for a ventilator,
* Having a congenital and genetic anomaly,
* Use of analgesic / Narcotic analgesic drugs,
* The mother has any substance abuse,
* Receiving continuous sedative therapy,
* Congenital malformation that can cause asphyxia and affect breathing
* Preterm newborns with intracranial hemorrhage formed the exclusion criteria of the study.

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile - PIPP | 1 year
  PIPP assesses pain with seven indicators. These are three behavioral (forehead wrinkles, enlargement of the eye wings and nose), two physiological (heart rate and oxygen saturation) and two contextual (gestational week and sleep/wake state) variables. The PIPP scale has 7 items to assess the baby's pain, such as gestational week, behavioral status, highest heart rate, lowest oxygen saturation value, forehead wrinkles, squint eyes, and enlarged nasal wings. Each item; It is scored from good to bad as 0, 1, 2, and 3. Premature Baby Pain Profile Scale is evaluated as mild pain between 0-6 points, moderate pain between 7-12 points and severe pain between 13-21 points.

SECONDARY OUTCOMES:
Heart Rate | 1 minute before the procedure. During the procedure. 1 minute and 2 minutes after the procedure
  The number of heartbeats per minute was obtained using an electrocardiographic bedside monitor and continuously recorded by custom computer software. An electrocardiographic bedside monitor was inserted into each of the infants.
Oxygen Saturation | 1 minute before the procedure. During the procedure. 1 minute and 2 minutes after the procedure
  Oxygen saturation (SpO2) was obtained using an electrocardiographic bedside monitor and continuously recorded by custom computer software. A separate an electrocardiographic bedside monitor was inserted into each of the infants.
Cerebral Oxygen Saturation (rScO2) | 1 minute before the procedure. During the procedure. 1 minute and 2 minutes after the procedure
  Cerebral Oxygen Saturation (rScO2) was obtained using an electrocardiographic bedside monitor and continuously recorded by custom computer software. A separate an electrocardiographic bedside monitor was inserted into each of the infants.
Measurement of incidence of adverse events | 1 minute before the procedure. During the procedure. 1 minute and 2 minutes after the procedure
  The safety of different interventions (Breast mılk pacıfıer, Sucrose pacıfıer and Pacıfıer) was assessed by the incidence of adverse events during the study period. The adverse events included: apnea, aspiration, cyanosis, tachycardia, bradycardia, tachypnea, dyspnea. The adverse events were monitored and recorded by specialist neonatal doctor who were blind to the purpose of the study. In case of a side effect, it was planned for the specialist neonatal doctor to stop the intervention immediately and to intervene.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK KONUKBAY, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University, Ankara
  - University of Health Sciences Turkey, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell-Yeo M, Johnston CC, Benoit B, Disher T, Caddell K, Vincer M, Walker CD, Latimer M, Streiner DL, Inglis D. Sustained efficacy of kangaroo care for repeated painful procedures over neonatal intensive care unit hospitalization: a single-blind randomized controlled trial. Pain. 2019 Nov;160(11):2580-2588. doi: 10.1097/j.pain.0000000000001646. PMID 31356452
- [Background] Chawanpaiboon S, Vogel JP, Moller AB, Lumbiganon P, Petzold M, Hogan D, Landoulsi S, Jampathong N, Kongwattanakul K, Laopaiboon M, Lewis C, Rattanakanokchai S, Teng DN, Thinkhamrop J, Watananirun K, Zhang J, Zhou W, Gulmezoglu AM. Global, regional, and national estimates of levels of preterm birth in 2014: a systematic review and modelling analysis. Lancet Glob Health. 2019 Jan;7(1):e37-e46. doi: 10.1016/S2214-109X(18)30451-0. Epub 2018 Oct 30. PMID 30389451
- [Background] Chen S, Zhang Q, Xie RH, Wen SW, Harrison D. What is the Best Pain Management During Gastric Tube Insertion for Infants Aged 0-12months: A Systematic Review. J Pediatr Nurs. 2017 May-Jun;34:78-83. doi: 10.1016/j.pedn.2016.12.015. Epub 2016 Dec 24. PMID 28024900
- [Background] Celik F, Sen S, Karayagiz Muslu G. Effects of Oral Stimulation and Supplemental Nursing System on the Transition Time to Full Breast of Mother and Sucking Success in Preterm Infants: A Randomized Controlled Trial. Clin Nurs Res. 2022 Jun;31(5):891-900. doi: 10.1177/10547738211058312. Epub 2021 Nov 16. PMID 34784787
- [Background] Fitri SYR, Lusmilasari L, Juffrie M, Bellieni CV. Modified Sensory Stimulation Using Breastmilk for Reducing Pain Intensity in Neonates in Indonesia: A Randomized Controlled Trial. J Pediatr Nurs. 2020 Jul-Aug;53:e199-e203. doi: 10.1016/j.pedn.2020.04.004. Epub 2020 May 10. PMID 32402558
- [Background] Ganguly A, Bhadesia PJ, Phatak AG, Nimbalkar AS, Nimbalkar SM. Pain profile of premature infants during routine procedures in neonatal intensive care: An observational study. J Family Med Prim Care. 2020 Mar 26;9(3):1517-1521. doi: 10.4103/jfmpc.jfmpc_1033_19. eCollection 2020 Mar. PMID 32509642
- [Background] Hoarau K, Payet ML, Zamidio L, Bonsante F, Iacobelli S. "Holding-Cuddling" and Sucrose for Pain Relief During Venepuncture in Newborn Infants: A Randomized, Controlled Trial (CASA). Front Pediatr. 2021 Jan 14;8:607900. doi: 10.3389/fped.2020.607900. eCollection 2020. PMID 33520895
- [Background] Kamity R, Kapavarapu PK, Chandel A. Feeding Problems and Long-Term Outcomes in Preterm Infants-A Systematic Approach to Evaluation and Management. Children (Basel). 2021 Dec 8;8(12):1158. doi: 10.3390/children8121158. PMID 34943354
- [Background] Li L, Wang L, Niu C, Liu C, Lv T, Ji F, Yu L, Yan W, Dou YL, Wang Y, Cao Y, Huang G, Hu X. Early skin contact combined with mother's breastfeeding to shorten the process of premature infants </= 30 weeks of gestation to achieve full oral feeding: the study protocol of a randomized controlled trial. Trials. 2021 Sep 17;22(1):637. doi: 10.1186/s13063-021-05605-x. PMID 34535164
- [Background] Lin T, Hu J, Zhang L, Qin X, Liu X, Lan Y, Chen K, You T. Promoting enteral tube feeding safety and performance in preterm infants: A systematic review. Int J Nurs Stud. 2022 Apr;128:104188. doi: 10.1016/j.ijnurstu.2022.104188. Epub 2022 Feb 4. PMID 35183863
- [Background] Mala O, Forster EM, Kain VJ. Neonatal Nurse and Midwife Competence Regarding Pain Management in Neonates: A Systematic Review. Adv Neonatal Care. 2022 Apr 1;22(2):E34-E42. doi: 10.1097/ANC.0000000000000911. Epub 2021 Jul 1. PMID 34224481
- [Background] McPherson C, Miller SP, El-Dib M, Massaro AN, Inder TE. The influence of pain, agitation, and their management on the immature brain. Pediatr Res. 2020 Aug;88(2):168-175. doi: 10.1038/s41390-019-0744-6. Epub 2020 Jan 2. PMID 31896130
- [Background] Mooney-Leber SM, Brummelte S. Neonatal pain and reduced maternal care: Early-life stressors interacting to impact brain and behavioral development. Neuroscience. 2017 Feb 7;342:21-36. doi: 10.1016/j.neuroscience.2016.05.001. Epub 2016 May 7. PMID 27167085
- [Background] Mooney-Leber SM, Brummelte S. Neonatal pain and reduced maternal care alter adult behavior and hypothalamic-pituitary-adrenal axis reactivity in a sex-specific manner. Dev Psychobiol. 2020 Jul;62(5):631-643. doi: 10.1002/dev.21941. Epub 2019 Dec 1. PMID 31788799
- [Background] Obeidat HM, Dwairej DA, Aloweidi AS. Pain in Preterm Infants: Different Perspectives. J Perinat Educ. 2021 Oct 1;30(4):185-195. doi: 10.1891/J-PE-D-20-00032. PMID 34908817
- [Background] Sener Taplak A, Erdem E. A Comparison of Breast Milk and Sucrose in Reducing Neonatal Pain During Eye Exam for Retinopathy of Prematurity. Breastfeed Med. 2017 Jun;12:305-310. doi: 10.1089/bfm.2016.0122. Epub 2017 Apr 17. PMID 28414522
- [Background] Velumula PK, Elbakoush F, Tabb C 2nd, Farooqi A, Lulic-Botica M, Jani S, Natarajan G, Bajaj M. Breast milk vs 24% sucrose for procedural pain relief in preterm neonates: a non-inferiority randomized controlled trial. J Perinatol. 2022 Jul;42(7):914-919. doi: 10.1038/s41372-022-01352-2. Epub 2022 Feb 23. PMID 35197549
- [Background] Williams MD, Lascelles BDX. Early Neonatal Pain-A Review of Clinical and Experimental Implications on Painful Conditions Later in Life. Front Pediatr. 2020 Feb 7;8:30. doi: 10.3389/fped.2020.00030. eCollection 2020. PMID 32117835
- [Background] Zhao T, Griffith T, Zhang Y, Li H, Hussain N, Lester B, Cong X. Early-life factors associated with neurobehavioral outcomes in preterm infants during NICU hospitalization. Pediatr Res. 2022 Dec;92(6):1695-1704. doi: 10.1038/s41390-022-02021-y. Epub 2022 Mar 25. PMID 35338349